CLINICAL TRIAL: NCT01143090
Title: A 24-Week, Flexible-Dose, Open-label Extension Study of Subjects Switched to Lurasidone for the Treatment of Schizophrenia or Schizoaffective Disorder (Protocol No. D1050290)
Brief Title: A Study of Subjects Switched to Lurasidone for the Treatment of Schizophrenia or Schizoaffective Disorder
Acronym: Switch Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050290
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Lurasidone; Latuda
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental): Subjects will continue on treatment with the same dose of lurasidone flexible dosing - 40 mg to 12 mg once daily taken orallay at endpoint of the D1050289 ( NCT01143077) core study.
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — 40 mg Lurasidone tablets, 40 - 120 mg per day for up to 6 months

SUMMARY:
Lurasidone (lurasidone HCl) is a novel psychotropic agent that is being developed as a potential new antipsychotic treatment for patients with schizophrenia. Switching between antipsychotic medications is common in the treatment of schizophrenia. The purpose of this study is to characterize the long-term safety and tolerability of lurasidone in subjects with schizophrenia or schizoaffective disorder and to allow for continued treatment for subjects completing the core study (D1050289-NCT01143077).

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed 6 weeks of treatment and all required assessments on the final study visit (Visit 8) of Study D1050289 (NCT01143077).

Exclusion Criteria:

* Subject is considered by the investigator to be at imminent risk of suicide or harm to self, others, or damage to property.
* Subject has a body mass index (BMI) greater than 40 or less than 18 kg/m2 (see Appendix 3 for BMI determination).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (27):
- United States (27):
  - K and S Professional Research Services, Little Rock, Arkansas
  - Synergy Clinical Research of Escondido, Escondido, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Pacific Research Partners, LLC, Oakland, California
  - California Clinical Trials, Paramount, California
  - Pasadena Research Institute, Pasadena, California
  - California Neuropsychopharmacology Clinical Research Institute (CNRI), LLC, Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Institute (CNRI), San Diego, California
  - University of California San Diego Medical Center, San Diego, California
  - Collaborative Neuroscience Network, South Bay, Torrance, California
  - Western Affiliated Research Institute, Denver, Colorado
  - Comprehensive NeuroScience, Inc., Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - St. Charles Psychiatric Associates - Midwest Research, Saint Charles, Missouri
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Duke University Dept. of Psychiatry, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - CRI Worldwide - Kirkbride Center, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Wharton Research Center, Wharton, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Result] Citrome L, Weiden PJ, McEvoy JP, Correll CU, Cucchiaro J, Hsu J, Loebel A. Effectiveness of lurasidone in schizophrenia or schizoaffective patients switched from other antipsychotics: a 6-month, open-label, extension study. CNS Spectr. 2014 Aug;19(4):330-9. doi: 10.1017/S109285291300093X. Epub 2013 Dec 16. PMID 24330868
- [Derived] Awad G, Ng-Mak D, Rajagopalan K, Hsu J, Pikalov A, Loebel A. Long-term health-related quality of life improvements among patients treated with lurasidone: results from the open-label extension of a switch trial in schizophrenia. BMC Psychiatry. 2016 Jun 1;16:176. doi: 10.1186/s12888-016-0879-5. PMID 27245981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FPI August 10, 2010-LPV November 28, 2011, locations were private health clinics, university hospitals, private research facilities.
Groups:
- Open Label: Subjects will continue on treatment with the same dose of lurasidone - 40 mg to 120 mg taken at endpoint of the D1050289 (NCT01143090) core study.
Period: Overall Study
Arm/Group | Open Label
Started | 149
Completed | 98
Not Completed | 51
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 17
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 18
Not completed — Non-compliance with study drug | 1
Not completed — Failure to meet eligibility criteria | 1
Not completed — Administrative | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label: Subjects will continue on treatment with the same dose of lurasidone - 40 mg to 120 mg taken at endpoint of the D1050289 (NCT01143090) core study. One enrolled subject did not receive any study medication and was excluded from this summary.
Arm/Group | Open Label
Number analyzed (Participants) | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 146
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 93
Region of Enrollment [Number; unit: participants] — One enrolled subject did not receive any study medication and was excluded from this summary.
  participants
    United States | 148

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Proportions of subjects with AEs, SAEs, and discontinuations due to AEs.
Time Frame: 6 months
Population: Safety population - One enrolled subject did not receive any study medication and was excluded from this summary.
Measure: Number; unit: participants
Arm/Group | Lurasidone Overall
Number analyzed (Participants) | 148
participants
  Any Treatment Emergent Adverse Event | 98
  Any Severe Treatment Emergent Adverse Event | 10
  Treatment Emergent AE Leading to Discontinuation | 16

2. Secondary Outcome: Efficacy
Description: Long-term efficacy of lurasidone in subjects with schizophrenia or schizoaffective disorder who have completed Study D1050289
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 8/148
Other Adverse Events (participants affected / at risk) | 47/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=148)
Schizoaffective Disorder (Psychiatric disorders) | 3 (3)
Schizophrenia (Psychiatric disorders) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 2 (2)
Bipolar I Disorder (Psychiatric disorders) | 1 (1)
Homicidal Ideation (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=148)
Nausea (Gastrointestinal disorders) | 13 (15)
Insomnia (Psychiatric disorders) | 13 (13)
Akathisia (Nervous system disorders) | 12 (12)
Anxiety (Psychiatric disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.